CLINICAL TRIAL: NCT06484023
Title: Place and Efficacy of Treatment With Posterior Tibial Transcutaneous Neurostimulation in Women With Idiopathic Overactive Bladder
Brief Title: Posterior Tibial Transcutaneous Neurostimulation in Idiopathic Overactive Bladder
Acronym: TENVESI
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-01
Record Dates: First submitted 2024-06-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Overactive Bladder
Keywords: neurostimulation
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Overactive bladder TENSI+ patients: Patients monitored for overactive bladder and using the TENSI + device for at least 3 months
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — quality of life questionnaire

SUMMARY:
Overactive bladder is a clinical diagnosis affecting up to 17% of women. The existing medical treatment, anticholinergics, has many side effects and is sometimes ineffective. Neurostimulation of the posterior tibial nerve is a validated 3rd-line therapy, after failure of perineal re-education and medication. Studies on TENS have shown a real impact on patients quality of life and encourage its use in routine clinical practice. TENSI+ medical device is a treatment for overactive bladder. It is non-invasive, placed over the posterior tibial nerve pathway and sends electrical stimulation via electrodes located on the skin. Discreet and without side effects for users, this treatment is indicated as 3rd-line treatment for people suffering from idiopathic overactive bladder with no contraindications. The aim of this study is to assess the quality of life of patients using this device, both before use and after at least 3 months of use.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for overactive bladder
* Patients using the TENSI+ for at least 3 months

Exclusion Criteria:

* Neurological disease that may explain overactive bladder
* Patient having received anticholinergic drug treatment during neurostimulation.
* Have one or more contraindications to wearing the device: pacemaker, defibrillator, wearing a mechanical implant near the electrode placement area, ankle joint problems, damaged skin, cognitive impairment.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients treated for overactive bladder and using the TENSI+ for at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Assessment of quality of life in patients who received treatment correctly treatment with TENSI + | Comparison before/after 3 month at least of TENS use
  Comparison of patients' quality of life with the OAB-q questionnaire after the installation of this therapy with patients' quality of life before the introduction of this therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No